CLINICAL TRIAL: NCT06577038
Title: Prospective, International, Multicenter, All-comers Registry for the Study of Intravascular Lithotripsy in Coronary Interventions
Brief Title: Prospective Registry on Intravascular Lithotripsy
Acronym: BENELUX-IVL
Status: Enrolling by invitation | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Principal Investigator, José M Montero Cabezas, Principal investigator, Leiden University Medical Center
Other Study IDs: CardioLUMC
Record Dates: First submitted 2024-07-22; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Calcific Coronary Arteriosclerosis
Keywords: calcific coronary lesions; intravascular lithotripsy; debulking; Complex percutaneous coronary interventions
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- IVL cohort: Patients with calcific CAD undergoing PCI and treated with IVL, irrespectively of the clinical indication (stable angina, acute coronary syndrome), anatomical scenario (de novo coronary stenosis, in-stent restenosis, etc) and/or concomitant use of other debulking techniques
  Interventions: Device: PCI with use of IVL

INTERVENTIONS:
Device: PCI with use of IVL — Use of IVL for the treatment of calcific coronary artery lesions at operator's discretion
  Other Names: Shockwave intravascular lithotripsy system

SUMMARY:
multicenter, international, all-comers registry aims to provide insights in the current application of IVL technology in patients with calcified coronary lesions undergoing PCI using IVL technology.

DETAILED DESCRIPTION:
The primary objectives are:

1. To analyze the trends of IVL use overall and according to clinical/anatomical indications
2. To evaluate the rates of procedural success, defined as success in facilitating stent delivery with <30% residual stenosis and without in-hospital
3. To describe the cumulative hierarchical incidence of MACE defined as: cardiac death, non-fatal target vessel myocardial infarction (MI), or clinically driven target lesion revascularization (TLR) at 30-days following the index procedure

The secondary objectives are:

1. To describe the rate of MACE at 3-, 6- and 12-months following the index procedure
2. To assess the rates of all causes mortality, clinically driven target lesion revascularization (TLR) or target vessel revascularization (TVR), any revascularization (non TLR, non TVR) and ARC-defined stent thrombosis at any time point, any type of angina at 30-days, 3-, 6- and 12-months following the index procedure
3. To describe the rates of target lesion failure (TLF) (see end-points definitions section)
4. To describe the rates of device crossing success (see end-points definitions section)
5. To describe the rates of serious angiographic complications (see end-points definitions section)
6. To assess predictors of clinical outcomes based on patient and procedural characteristics
7. To analyze current standards of practice regarding IVL technology in a real-world multinational cohort (technique, training, local protocols).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years-old
* Ability to provide written informed consent

Exclusion Criteria:

* Patient has any comorbidity or condition that, in the opinion of the Investigator, compromises the subject's ability to give written informed consent
* Patient belongs to a vulnerable population Subject is a member of a vulnerable population , including individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with calcific CAD undergoing PCI and treated with IVL, irrespectively of the clinical indication (stable angina, acute coronary syndrome), anatomical scenario (de novo coronary stenosis, in-stent restenosis due to poorly stent expansion) and/or concomitant use of other debulking techniques (e.g. RA).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
procedural success | Periprocedurally and from hospital admission to discharge (an average of 2 days)
  success in facilitating stent delivery with <30% residual stenosis and without in-hospital MACE
cumulative hierarchical incidence of MACE | At 30 days follow-up
  cardiac death, non-fatal target vessel myocardial infarction (MI), or clinically driven target lesion revascularization (TLR) at 30-days following the index procedure

SECONDARY OUTCOMES:
rate of MACE at 3 months | At 3 months follow-up
  rate of MACE at 3-months following the index procedure
rate of MACE at 6 months | At 6 months follow-up
  rate of MACE at 6-months following the index procedure
rate of MACE at 12 months | At 12 months follow-up
  rate of MACE at 12-months following the index procedure
the rates of all causes mortality, clinically driven target lesion revascularization (TLR) or target vessel revascularization (TVR), any revascularization (non TLR, non TVR) and ARC-defined stent thrombosis | 30-days, 3-, 6- and 12-months
  at any time point, any type of angina at 30-days, 3-, 6- and 12-months following the index procedure
the rates of all causes mortality, clinically driven target lesion revascularization (TLR) or target vessel revascularization (TVR), any revascularization (non TLR, non TVR) and ARC-defined stent thrombosis | at 30-days follow-up
  at any time point, any type of angina at 30-days follow-up
the rates of all causes mortality, clinically driven target lesion revascularization (TLR) or target vessel revascularization (TVR), any revascularization (non TLR, non TVR) and ARC-defined stent thrombosis | at 3 months follow-up
  at any time point, any type of angina at 3 months follow-up
the rates of all causes mortality, clinically driven target lesion revascularization (TLR) or target vessel revascularization (TVR), any revascularization (non TLR, non TVR) and ARC-defined stent thrombosis | at 6 months follow-up
  at any time point, any type of angina at 6 months follow-up
the rates of all causes mortality, clinically driven target lesion revascularization (TLR) or target vessel revascularization (TVR), any revascularization (non TLR, non TVR) and ARC-defined stent thrombosis | at 12-months follow-up
  at any time point, any type of angina at 12-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: José M Montero Cabezas, MD PhD, Study Chair — Leiden University Medical Center; Ibtihal Al Amri, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (8):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Red Cross Hospital, Athens, Greece
- Netherlands (6):
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Rijnstate Ziekenhuis, Arnhem
  - Medisch Centrum Leeuwaarden, Leeuwarden
  - Radboud University Medical Center, Nijmegen

REFERENCES:
- [Background] Kawashima H, Serruys PW, Hara H, Ono M, Gao C, Wang R, Garg S, Sharif F, de Winter RJ, Mack MJ, Holmes DR, Morice MC, Kappetein AP, Thuijs DJFM, Milojevic M, Noack T, Mohr FW, Davierwala PM, Onuma Y; SYNTAX Extended Survival Investigators. 10-Year All-Cause Mortality Following Percutaneous or Surgical Revascularization in Patients With Heavy Calcification. JACC Cardiovasc Interv. 2022 Jan 24;15(2):193-204. doi: 10.1016/j.jcin.2021.10.026. Epub 2021 Dec 29. PMID 34973904
- [Background] Rheude T, Koch T, Joner M, Lenz T, Xhepa E, Wiebe J, Coughlan JJ, Aytekin A, Cassese S, Laugwitz KL, Schunkert H, Kastrati A, Kufner S. Ten-year clinical outcomes of drug-eluting stents with different polymer coating strategies by degree of coronary calcification: a pooled analysis of the ISAR-TEST 4 and 5 randomised trials. EuroIntervention. 2023 Feb 20;18(14):1188-1196. doi: 10.4244/EIJ-D-22-00781. PMID 36453826
- [Background] Lee MS, Shah N. The Impact and Pathophysiologic Consequences of Coronary Artery Calcium Deposition in Percutaneous Coronary Interventions. J Invasive Cardiol. 2016 Apr;28(4):160-7. Epub 2015 Aug 25. PMID 26301561
- [Background] Madhavan MV, Tarigopula M, Mintz GS, Maehara A, Stone GW, Genereux P. Coronary artery calcification: pathogenesis and prognostic implications. J Am Coll Cardiol. 2014 May 6;63(17):1703-14. doi: 10.1016/j.jacc.2014.01.017. Epub 2014 Feb 12. PMID 24530667
- [Background] Mintz GS. Intravascular imaging of coronary calcification and its clinical implications. JACC Cardiovasc Imaging. 2015 Apr;8(4):461-471. doi: 10.1016/j.jcmg.2015.02.003. PMID 25882575
- [Background] Kassimis G, Raina T, Kontogiannis N, Patri G, Abramik J, Zaphiriou A, Banning AP. How Should We Treat Heavily Calcified Coronary Artery Disease in Contemporary Practice? From Atherectomy to Intravascular Lithotripsy. Cardiovasc Revasc Med. 2019 Dec;20(12):1172-1183. doi: 10.1016/j.carrev.2019.01.010. Epub 2019 Jan 10. PMID 30711477
- [Background] Barbato E, Gallinoro E, Abdel-Wahab M, Andreini D, Carrie D, Di Mario C, Dudek D, Escaned J, Fajadet J, Guagliumi G, Hill J, McEntegart M, Mashayekhi K, Mezilis N, Onuma Y, Reczuch K, Shlofmitz R, Stefanini G, Tarantini G, Toth GG, Vaquerizo B, Wijns W, Ribichini FL. Management strategies for heavily calcified coronary stenoses: an EAPCI clinical consensus statement in collaboration with the EURO4C-PCR group. Eur Heart J. 2023 Nov 1;44(41):4340-4356. doi: 10.1093/eurheartj/ehad342. PMID 37208199
- [Background] Hill JM, Kereiakes DJ, Shlofmitz RA, Klein AJ, Riley RF, Price MJ, Herrmann HC, Bachinsky W, Waksman R, Stone GW; Disrupt CAD III Investigators. Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Artery Disease. J Am Coll Cardiol. 2020 Dec 1;76(22):2635-2646. doi: 10.1016/j.jacc.2020.09.603. Epub 2020 Oct 15. PMID 33069849
- [Background] Forero MNT, Daemen J. The Coronary Intravascular Lithotripsy System. Interv Cardiol. 2019 Nov 18;14(3):174-181. doi: 10.15420/icr.2019.18.R1. eCollection 2019 Nov. PMID 31867065
- [Background] Kereiakes DJ, Di Mario C, Riley RF, Fajadet J, Shlofmitz RA, Saito S, Ali ZA, Klein AJ, Price MJ, Hill JM, Stone GW. Intravascular Lithotripsy for Treatment of Calcified Coronary Lesions: Patient-Level Pooled Analysis of the Disrupt CAD Studies. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1337-1348. doi: 10.1016/j.jcin.2021.04.015. Epub 2021 May 3. PMID 33939604
- [Background] Ali ZA, Brinton TJ, Hill JM, Maehara A, Matsumura M, Karimi Galougahi K, Illindala U, Gotberg M, Whitbourn R, Van Mieghem N, Meredith IT, Di Mario C, Fajadet J. Optical Coherence Tomography Characterization of Coronary Lithoplasty for Treatment of Calcified Lesions: First Description. JACC Cardiovasc Imaging. 2017 Aug;10(8):897-906. doi: 10.1016/j.jcmg.2017.05.012. PMID 28797412
- [Background] Sianos G, Morel MA, Kappetein AP, Morice MC, Colombo A, Dawkins K, van den Brand M, Van Dyck N, Russell ME, Mohr FW, Serruys PW. The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease. EuroIntervention. 2005 Aug;1(2):219-27. No abstract available. PMID 19758907
- [Background] Mintz GS, Popma JJ, Pichard AD, Kent KM, Satler LF, Chuang YC, Ditrano CJ, Leon MB. Patterns of calcification in coronary artery disease. A statistical analysis of intravascular ultrasound and coronary angiography in 1155 lesions. Circulation. 1995 Apr 1;91(7):1959-65. doi: 10.1161/01.cir.91.7.1959. PMID 7895353
- [Background] Tearney GJ, Regar E, Akasaka T, Adriaenssens T, Barlis P, Bezerra HG, Bouma B, Bruining N, Cho JM, Chowdhary S, Costa MA, de Silva R, Dijkstra J, Di Mario C, Dudek D, Falk E, Feldman MD, Fitzgerald P, Garcia-Garcia HM, Gonzalo N, Granada JF, Guagliumi G, Holm NR, Honda Y, Ikeno F, Kawasaki M, Kochman J, Koltowski L, Kubo T, Kume T, Kyono H, Lam CC, Lamouche G, Lee DP, Leon MB, Maehara A, Manfrini O, Mintz GS, Mizuno K, Morel MA, Nadkarni S, Okura H, Otake H, Pietrasik A, Prati F, Raber L, Radu MD, Rieber J, Riga M, Rollins A, Rosenberg M, Sirbu V, Serruys PW, Shimada K, Shinke T, Shite J, Siegel E, Sonoda S, Suter M, Takarada S, Tanaka A, Terashima M, Thim T, Uemura S, Ughi GJ, van Beusekom HM, van der Steen AF, van Es GA, van Soest G, Virmani R, Waxman S, Weissman NJ, Weisz G; International Working Group for Intravascular Optical Coherence Tomography (IWG-IVOCT). Consensus standards for acquisition, measurement, and reporting of intravascular optical coherence tomography studies: a report from the International Working Group for Intravascular Optical Coherence Tomography Standardization and Validation. J Am Coll Cardiol. 2012 Mar 20;59(12):1058-72. doi: 10.1016/j.jacc.2011.09.079. Erratum In: J Am Coll Cardiol. 2012 May 1;59(18):1662. Dudeck, Darius [corrected to Dudek, Darius]; Falk, Erlin [corrected to Falk, Erling]; Garcia, Hector [corrected to Garcia-Garcia, Hector M]; Sonada, Shinjo [corrected to Sonoda, Shinjo]; Troels, Thim [corrected to Thim, Troels]; van Es, Gerrit-Ann [correct. PMID 22421299
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Bass TA. High-Risk Percutaneous Coronary Interventions in Modern Day Clinical Practice: Current Concepts and Challenges. Circ Cardiovasc Interv. 2015 Dec;8(12):e003405. doi: 10.1161/CIRCINTERVENTIONS.115.003405. No abstract available. PMID 26628592
- [Background] Saito S, Yamazaki S, Takahashi A, Namiki A, Kawasaki T, Otsuji S, Nakamura S, Shibata Y; Disrupt CAD IV Investigators. Intravascular Lithotripsy for Vessel Preparation in Calcified Coronary Arteries Prior to Stent Placement - Japanese Disrupt CAD IV Study 1-Year Results. Circ Rep. 2022 Aug 20;4(9):399-404. doi: 10.1253/circrep.CR-22-0068. eCollection 2022 Sep 9. PMID 36120480
- [Background] Abdel-Wahab M, Richardt G, Joachim Buttner H, Toelg R, Geist V, Meinertz T, Schofer J, King L, Neumann FJ, Khattab AA. High-speed rotational atherectomy before paclitaxel-eluting stent implantation in complex calcified coronary lesions: the randomized ROTAXUS (Rotational Atherectomy Prior to Taxus Stent Treatment for Complex Native Coronary Artery Disease) trial. JACC Cardiovasc Interv. 2013 Jan;6(1):10-9. doi: 10.1016/j.jcin.2012.07.017. Epub 2012 Dec 19. PMID 23266232
- [Background] Sardella G, Stefanini G, Leone PP, Boccuzzi G, Fovero NT, Van Mieghem N, Giacchi G, Escaned J, Fineschi M, Testa L, Valenti R, Di Mario C, Briguori C, Cortese B, Ribichini F, Oreglia JA, Colombo A, Sangiorgi G, Barbato E, Sonck J, Ugo F, Trani C, Castriota F, Paggi A, Porto I, Tomai F, Mancone M. Coronary Lithotripsy as Elective or Bail-Out Strategy After Rotational Atherectomy in the Rota-Shock Registry. Am J Cardiol. 2023 Jul 1;198:1-8. doi: 10.1016/j.amjcard.2023.04.032. Epub 2023 May 12. PMID 37182254
- [Background] Mousa MAA, Bingen BO, Al Amri I, Mertens BJA, Taha S, Tohamy A, Youssef A, Jukema JW, Montero-Cabezas JM. Efficacy and Safety of Intravascular Lithotripsy Versus Rotational Atherectomy in Balloon-Crossable Heavily Calcified Coronary Lesions. Cardiovasc Revasc Med. 2023 Mar;48:1-6. doi: 10.1016/j.carrev.2022.10.011. Epub 2022 Oct 29. No abstract available. PMID 36336588
- [Background] Rodriguez-Leor O, Cid-Alvarez AB, Lopez-Benito M, Gonzalo N, Vilalta V, Diarte de Miguel JA, Lopez LF, Jurado-Roman A, Diego A, Oteo JF, Cuellas C, Trillo R, Travieso A, Alfonso F, Carrillo X, Vegas-Valle JM, Cortes-Villar C, Pascual I, Munoz Camacho JF, Flores X, Vera-Vera S, Moreu J, Barreira de Sousa G, Marti D, Jimenez-Mazuecos J, Fuertes M, Ocaranza R, de la Torre Hernandez JM, Lozano F, Solana Martinez SG, Gomez-Lara J, Perez de Prado A; REPLICA-EPIC18 Investigators. A Prospective, Multicenter, Real-World Registry of Coronary Lithotripsy in Calcified Coronary Arteries: The REPLICA-EPIC18 Study. JACC Cardiovasc Interv. 2024 Mar 25;17(6):756-767. doi: 10.1016/j.jcin.2023.12.018. Epub 2024 Feb 21. PMID 38385926
- [Derived] Oliveri F, Garcia PV, van Oort MJH, Phagu A, Al Amri I, Bingen BO, Paradies V, Mincione G, Claessen BE, Dimitriu-Leen AC, Kefer J, Girgis H, Vossenberg T, Mandurino-Mirizzi A, Van der Kley F, Jukema JW, Montero-Cabezas JM. Intravascular lithotripsy for the treatment of calcified coronary lesions in individuals of advanced age: a post-hoc analysis of the multicentre, prospective BENELUX-IVL study. EClinicalMedicine. 2025 Jul 4;85:103342. doi: 10.1016/j.eclinm.2025.103342. eCollection 2025 Jul. PMID 40686682
- [Derived] van Oort MJH, Bingen BO, Oliveri F, Al Amri I, Phagu AAS, Claessen BEPM, Dimitriu-Leen AC, Vossenberg TN, Kefer J, Girgis H, van der Kley F, Jukema JW, Montero-Cabezas JM. Clinical and Technical Predictors of Treatment Success After Coronary Intravascular Lithotripsy in Calcific Coronary Lesions. Catheter Cardiovasc Interv. 2025 May;105(6):1418-1426. doi: 10.1002/ccd.31480. Epub 2025 Mar 4. PMID 40038885